CLINICAL TRIAL: NCT06639529
Title: Preliminary Study of CXCL3 As a Biomarker of Diabetic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-695
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Kidney Disease (DKD)
Keywords: CXCL3; biomarker; urine; serum; renal tissue
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- normal control (Experimental): Tests of the expression of CXCL3 in various tissues
  Interventions: Diagnostic Test: Tests of the expression of CXCL3 in various tissues
- diabetic mellitus (Experimental): Tests of the expression of CXCL3 in various tissues
  Interventions: Diagnostic Test: Tests of the expression of CXCL3 in various tissues
- diabetic kidney disease (Experimental): Tests of the expression of CXCL3 in various tissues
  Interventions: Diagnostic Test: Tests of the expression of CXCL3 in various tissues

INTERVENTIONS:
Diagnostic Test: Tests of the expression of CXCL3 in various tissues — 1.The expression of CXCL3 in peripheral blood PBMC was detected by RT-qPCR. 2.The levels of CXCL3 in serum and urine were detected by Elisa method. 3.Clinical data collection includes the patient 's name, gender, weight, height, biochemical indicators, urine test indicators, renal biopsy data, etc. 4.The expression of CXCL3 in renal tissue was determined by immunohistochemistry.

SUMMARY:
The goal of this study is to learn about CXCL3 as a biomarker for type 2 diabetic kidney disease (DKD) in adults between age of 18-80. The main question it aims to answer is:

* Is CXCL3 elevated in the serum or urine of type 2 adult DKD patients compared to normal control or diabetes mellitus without kidney involvement?
* Is CXCL3 elevated in the mRNA of PBMC of type 2 adult DKD patients compared to normal control or diabetes mellitus without kidney involvement?
* Is CXCL3 elevated in the kidney tissue of type 2 adult DKD patients compared to normal control or other glomerulonephritis? Participants have already been diagnosed as DKD by renal biopsy.

DETAILED DESCRIPTION:
Diabetic kidney disease ( DKD ) has become the first cause of end-stage renal disease. The high cost of treatment brings a heavy burden to the social economy and medical insurance. However, the pathogenesis of DKD is still unclear. Because the early symptoms of DKD are hidden and difficult to diagnose, once a large amount of proteinuria occurs in clinical practice, renal damage is often difficult to reverse, and patients will soon enter ESRD. Therefore, it is of great social significance and economic benefits to clarify the pathogenesis of DKD and find more effective therapeutic targets for DKD.In our previous bioinformatics analysis, it was found that CXCL3 was significantly increased in peripheral blood PBMC of DKD, and CXCL3 was the core gene of DKD after screening by WGCNA and machine learning. CXC legend 3 ( CXCL3 ), also known as GRO gamma ( GROγ ), is a 7.9 kDa protein composed of 73 amino acids. CXCL3 is a member of the CXC subfamily of chemokines, including the ' ELR ' motif of its receptor CXCR2 tuberculosis. CXCL3 is considered to be a chemotactic factor for neutrophils, while CXCL3 has other proven roles in the field of cancer. Studies have shown that serum CXCL3 levels are associated with the progression and poor prognosis of colorectal cancer, and CXCL3 overexpression increases the malignant behavior of tumor cells, while down-regulation of its expression inhibits this phenomenon. The CXCL3 released by macrophages can promote the transformation of fibroblasts into myofibroblasts, thereby promoting the metastasis of pancreatic cancer. However, there are still few studies on CXCL3 in the kidney, and its role in DKD needs to be further explored. In the DKD single cell dataset and the KIT website, we found that CXCL3 was significantly increased in DKD, and was positively correlated with proteinuria and serum creatinine. On the basis of previous bioinformatics analysis and verification, this study further verified that the gene had no DKD damage in DKD and diabetes, the mRNA expression level of peripheral blood PBMC in normal control and the expression level in serum and urine ( Elisa ), and further verified in kidney tissue, animal and cell levels, looking for new biomarkers for DKD.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical and pathological diagnosis of diabetic kidney disease;
* 2. Clinical diagnosis of type 2 diabetes mellitus.

Exclusion Criteria:

* 1. Tumor;
* 2. Active infection;
* 3. Heart failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Serum and Urine CXCL3 level by Enzyme linked immunosorbent assay (Elisa) | From enrollment to the end of experiment at 4 weeks
  Serum and Urine samples were thawed and subjected to centrifugation. Thereafter, the levels of CXCL3 were determined using a sandwich ELISA kit.

SECONDARY OUTCOMES:
Immunohistochemistry and immunofluorescence of CXCL3 in kidney tissue | From enrollment to the end of experiment at 8 weeks
  The kidney tissues of DKD patients and normal/disease controls were fixed in formalin and then paraffin-embedded to prepare renal sections. The prepared renal section was stained with CXCL3 antibody, and images were captured using an Olympus cellSens Entry microscopy system.

OTHER OUTCOMES:
mRNA level of CXCL3 in PBMC | From enrollment to the end of experiment at 4 weeks
  Total RNA was isolated from these cells using a Total RNA Isolation Kit, RT-qPCR of PBMC in DKD and normal controls was conducted using 2× Q3 SYBR qPCR Master mix.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No
The primary concern is the protection of participant privacy. Even with anonymization techniques, there is a risk of re-identification, particularly in studies involving rare diseases or specific populations. Participants trust researchers to safeguard their personal information, and any breach of this trust could have serious implications for their well-being. Maintaining confidentiality is not only an ethical obligation but also a legal one, as regulations such as the Health Insurance Portability and Accountability Act (HIPAA) in the United States mandate strict guidelines for handling sensitive health information.
  Sharing individual participant data without proper context can lead to misinterpretation and misuse of the data. Researchers or stakeholders who are not involved in the study may draw erroneous conclusions or apply the findings inappropriately. This misinterpretation can undermine the credibility of the research and could potentially lead to harmful consequences for patien